CLINICAL TRIAL: NCT05929794
Title: Impact of Formulation on the Pharmacokinetics of Micropatch-assisted Delivery of Metronidazole
Brief Title: Pharmacokinetics of Transdermal Metronidazole
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Nicole K Brogden, Associate Professor, University of Iowa
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202211064
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Microneedle; Micropatch; Transdermal; Metronidazole
MeSH Terms: interventions — Metronidazole; Gels; Electric Impedance

STUDY DESIGN:
Intervention Model Description: This is an open-label, 2-way crossover, non-placebo controlled pharmacokinetic assessment study in n=24 health adult subjects. In this crossover study, all subjects will receive treatment with either metronidazole gel or cream, depending on assigned study group. During different periods of the study, the metronidazole product will be applied to skin treated with a micropatch (period 1) and to skin not treated with a micropatch (period 2) on the upper arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Micropatch application + metronidazole 0.75% topical gel (Active Comparator): Participants will have pre-treatment micropatch application followed by metronidazole 0.75% topical gel
  Interventions: Drug: Metronidazole 0.75% Topical Gel; Diagnostic Test: Transdermal water loss measurement; Diagnostic Test: Electrical Resistance; Diagnostic Test: Skin color measurement; Other: Micropatch application
- Metronidazole 0.75% topical gel (Active Comparator): Participants will have metronidazole 0.75% topical gel applied without the pre-treatment micropatch application
  Interventions: Drug: Metronidazole 0.75% Topical Gel; Diagnostic Test: Transdermal water loss measurement; Diagnostic Test: Electrical Resistance; Diagnostic Test: Skin color measurement
- Micropatch application + metronidazole 0.75% topical cream (Active Comparator): Participants will have pre-treatment micropatch application followed by metronidazole 0.75% topical cream
  Interventions: Drug: Metronidazole 0.75% Topical Cream; Diagnostic Test: Transdermal water loss measurement; Diagnostic Test: Electrical Resistance; Diagnostic Test: Skin color measurement; Other: Micropatch application
- Metronidazole 0.75% topical cream (Active Comparator): Participants will have metronidazole 0.75% topical cream applied without the pre-treatment micropatch application
  Interventions: Drug: Metronidazole 0.75% Topical Cream; Diagnostic Test: Transdermal water loss measurement; Diagnostic Test: Electrical Resistance; Diagnostic Test: Skin color measurement

INTERVENTIONS:
Drug: Metronidazole 0.75% Topical Gel — Half of enrolled subjects will undergo this intervention. Baseline measurements of transepidermal water loss, electrical resistance, and color will be made at 3 sites on the upper arm. Color will only be measured at baseline. Micropatch application will occur at 2 sites, followed by application of metronidazole gel and then covered with an occlusive covering. One site will be covered with an occlusive covering only (no micropatch or gel). At 48 hours occlusive coverings and gel are removed and electrical resistance measurements are repeated. Fresh gel and occlusive patches are reapplied. At 96 hours the patches are removed and electrical resistance measurements repeated. Blood samples are taken daily for 5 days. Measurements from the 3rd site allow each subject to serve as their own control in data analysis. After a minimum 7 days washout period, all of these procedures will be repeated again except that there will be no micropatch application at any of the 3 sites.
  Arms: Metronidazole 0.75% topical gel; Micropatch application + metronidazole 0.75% topical gel
Drug: Metronidazole 0.75% Topical Cream — Half of enrolled subjects will undergo this intervention. Baseline measurements of transepidermal water loss, electrical resistance, and color will be made at 3 sites on the upper arm. Color will only be measured at baseline. Micropatch application will occur at 2 sites, followed by application of metronidazole cream and then covered with an occlusive covering. One site will be covered with an occlusive covering only (no micropatch or cream). At 48 hours occlusive coverings and cream are removed and electrical resistance measurements are repeated. Fresh cream and occlusive patches are reapplied. At 96 hours the patches are removed and electrical resistance measurements repeated. Blood samples are taken daily for 5 days. Measurements from the 3rd site allow each subject to serve as their own control in data analysis. After a minimum 7 days washout period, all of these procedures will be repeated again except that there will be no micropatch application at any of the 3 sites.
  Arms: Metronidazole 0.75% topical cream; Micropatch application + metronidazole 0.75% topical cream
Diagnostic Test: Transdermal water loss measurement — Baseline measurements of transepidermal water loss will be made at 3 sites on the upper arm. In the study periods that have micropatch application, the measurements will be repeated after micropatch application and removal (before any metronidazole product is applied).
Diagnostic Test: Electrical Resistance — Baseline measurements of electrical resistance will be made at 3 sites on the upper arm. In the study periods that have micropatch application, the measurements will be repeated after micropatch application and removal (before any metronidazole product is applied). In all study periods the measurements will also be repeated at 48 hours and 96 hours, when metronidazole product and occlusive coverings are removed from the skin.
Diagnostic Test: Skin color measurement — Baseline measurements of skin color will be made at 3 sites on the upper arm.
Other: Micropatch application — All subjects will undergo this intervention. Baseline measurements of transepidermal water loss, electrical resistance, and color will be made at 3 sites on the upper arm (color only measured at baseline). Two sites will have micropatch application + metronidazole product with occlusive covering. One site will have micropatch application + occlusive covering, no metronidazole product. Micropatch application will only occur on day 1 (a micropatch is a patch of 50 microneedles). Transepidermal water loss and electrical resistance are repeated after micropatch application and removal. At 48 hours occlusive coverings and metronidazole are removed; electrical resistance measurements are repeated. Metronidazole product and fresh occlusive patches are reapplied. At 96 hours patches are removed and electrical resistance measurements repeated. Blood samples are taken daily for 5 days. Measurements from the 3rd site allow each subject to serve as their own control in data analysis.
  Arms: Micropatch application + metronidazole 0.75% topical cream; Micropatch application + metronidazole 0.75% topical gel

SUMMARY:
This is a crossover pharmacokinetic clinical study in healthy volunteers to compare metronidazole delivery through skin when a gel or cream metronidazole product is applied to skin treated with a micropatch.

DETAILED DESCRIPTION:
The goal of this crossover pharmacokinetic clinical study in healthy volunteers is to compare metronidazole delivery through skin when a gel or cream metronidazole product is applied to skin treated with a micropatch. The main questions this study aims to answer are:

* Is micropatch transdermal delivery dependent on the metronidazole product formulation?
* Is transdermal delivery dependent on micropore lifetime of the skin after micropatch application?

Participants will be divided into groups based on metronidazole product (gel or cream).

* The metronidazole product will be applied to micropatch-treated skin in study period one. Measurements of the skin barrier will be made before and after micropatch treatment.
* Daily blood samples will be collected for up to 5 days after the micropatch and metronidazole are first applied.
* Following a one-week washout period, the same study process will be repeated except that metronidazole product will be applied to skin without micropatch pretreatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women ≥18 years old, of any ethnic background
* Provide written informed consent before initiation of any study procedures
* Available for follow-up for the planned duration of the study
* Able to communicate well with the investigators
* Able to adhere to the study protocol schedule, study restrictions and examination schedule
* Subjects deemed to be healthy, as determined by the study physician, based on medical history, current medical conditions, and medication history
* Agrees not to participate in another clinical study during the study period unless the study is in the follow up phase and it has been 1 month since the subject received any experimental agents or treatments. The subject also agrees not to participate in an investigational drug study for at least 1 month after last procedure day
* Agrees not to donate blood to a blood bank throughout participation in the study and for at least 2 months after last procedure day.

Exclusion Criteria:

* Unable to give consent
* Inability to communicate or cooperate with the investigators
* Known previous adverse reaction to microneedle insertion
* Known allergy or adverse reaction to medical tape/adhesive, or aloe vera
* Women who are pregnant or lactating
* Abnormal vital signs or lab values deemed to be medically significant by the study physician or Principal Investigator
* Positive urine drug screening test
* Known prior serious adverse reaction or hypersensitivity to metronidazole or any metronidazole products
* History of anaphylaxis to an antibiotic, antimicrobial, antifungal, antipartisitic, or antiviral drug
* Current smoker or regular use of nicotine or tobacco products
* Participation in any ongoing investigational drug trial or clinical drug trial unless the study is in the follow up phase and it has been ≥1 month since the subject received any experimental agents or treatments
* Current use of medications in the following therapeutic classes: HMGCoA reductase inhibitors ("statins"), beta-blockers, oral or topical steroids, oral antibiotics, topical antibiotics at the local treatment site, topical antihistamines at the local treatment site, and oral or topical NSAIDs/analgesics. A subject who has recently used oral or topical steroids, antibiotics, antihistamines, or NSAIDs/analgesics may be enrolled if more than 5 elimination half-lives of the drug have passed since the last dose. The estimated elimination half-life for any specific drug will be obtained from standard pharmacy references such as Micromedex or other comparable references.
* Current or recent use of any prescription medication that, in the opinion of the study physician or Principal Investigator, would present a safety risk when used concomitantly with metronidazole
* Any current medical conditions (acute or chronic) that may pose a risk for study participation, as determined by the study physician or Principal Investigator
* Any condition that would, in the opinion of the study physician or Principal Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
* Uncontrolled mental illness that would, in the opinion of the study physician or Principal Investigator, affect the subject's ability to understand or reliably participate in the study
* Subject has presence of a skin condition, excessive hair at the application site, sunburn, raised moles and scars, open sores at application site, scar tissue, tattoo, coloration, or any other local condition that would interfere with placement of patches, microneedles, study drug, skin assessment, or reactions to drug
* Medical history of significant dermatologic diseases or conditions, such as atopy, psoriasis, vitiligo or conditions known to alter skin appearance or physiologic response (e.g. diabetes, porphyria).
* Any current malignancy or history of malignancy at the treatment site
* Prior history of keloids or excessive scarring
* Prior history of skin pigmentation changes or significant dermal reaction to a topically applied drug product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of maximum serum metronidazole concentration (Cmax) | 0.5, 1, 1.5, 2, 4, 6, 8, 24, 48, 72, 96, 98, 100, 104, and 120 hours
  Cmax is the highest metronidazole concentration measured in the serum.
Time of maximum serum metronidazole concentration (Tmax) | 0.5, 1, 1.5, 2, 4, 6, 8, 24, 48, 72, 96, 98, 100, 104, and 120 hours
  Tmax is the time point at which the maximum drug concentration in serum is measured.
Area under the serum-concentration curve from 0-120 hours | 0.5, 1, 1.5, 2, 4, 6, 8, 24, 48, 72, 96, 98, 100, 104, and 120 hours
  Area under the serum-concentration-time curve is a mathematical measure of total systemic exposure to metronidazole in the body.

SECONDARY OUTCOMES:
Skin color | Baseline (Day 1)
  Lightness/darkness of the skin is measured with a tristimulus colorimeter and reported in a unitless value called L*. Higher L* values denote lighter skin, while lower L* values denote darker skin. Data are collected as the mean of measurements from 3 sites on the upper arm.
Change in transepidermal water loss after micropatch application | Baseline (Day 1) and post-micropatch application (Day 1)
  The percent change in transepidermal water loss from baseline to post-micropatch application at the upper arm sites will be calculated. These data are only collected from the micropatch sites. Percent change is calculated as (transepidermal water loss after micropatch application/baseline transepidermal water loss) x 100. Data will be calculated as the mean of measurements from micropatch application sites at the upper arm.
Change in electrical resistance after micropatch application | Baseline (Day 1) and post-micropatch application (Day 1)
  The percent change in electrical resistance from baseline to post-micropatch application at the upper arm sites will be calculated. These data are only collected from the micropatch sites. Percent change is calculated as (electrical resistance after micropatch application/baseline electrical resistance) x 100. Data will be calculated as the mean of measurements from micropatch application sites at the upper arm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No